CLINICAL TRIAL: NCT03946735
Title: Cognitive Behavioural Therapy as an Effective Treatment for Social Anxiety, Perfectionism, and Rumination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alzahra University (Other)
Responsible Party: Principal Investigator, Abbas Abdollahi, Principal investigator, Alzahra University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alzahra123456789
Record Dates: First submitted 2019-05-07; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety; Perfectionism; Rumination; Cognitive Behavioural Therapy
MeSH Terms: conditions — Phobia, Social; Rumination Syndrome | interventions — Cognitive Behavioral Therapy; Rumination, Digestive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention study (Experimental): Cognitive Behavioural Therapy for social anxiety
  Interventions: Behavioral: Cognitive Behavioural Therapy as an Effective Treatment for Social Anxiety, Perfectionism, and Rumination
- Social anxiety (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Therapy as an Effective Treatment for Social Anxiety, Perfectionism, and Rumination

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy as an Effective Treatment for Social Anxiety, Perfectionism, and Rumination — Week one involved introducing CBT and assessing the negative effects of perfectionism, rumination, and social anxiety. Week two allowed participants to specify stressful social activities, stressful social situations, and enjoyable activities. Week three to week six allowed participants to identify automatic thoughts and thinking errors (for example, all or nothing thinking, self-criticism, dysfunctional schemas for self-evaluation, and unrealistic standards). Assignments were provided to participants with the content of exposure to anxiety evoking situations in the treatment sessions and at home. Achievable behavioural goals were set for participants in the treatment sessions and at home.

SUMMARY:
This randomized, controlled trial study was designed to examine the efficacy of Cognitive Behavioural Therapy (CBT) on social anxiety, perfectionism, and rumination among individuals diagnosed with social anxiety in Tehran, Iran.

DETAILED DESCRIPTION:
A total of 52 individuals with Social Anxiety Disorder (SAD) (68% female, mean age = 35.67) were allocated to a CBT group or to a control group. The intervention group was given one session of therapy per week over a duration of 8 weeks, while the control group did not receive any intervention and was placed on a waiting list. Self-reported social anxiety, perfectionism, and rumination were measured before the CBT intervention, after the intervention, and two months after the intervention for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants formally diagnosed with SAD by psychologists who determined the individual meet criteria outlined by the Diagnostic and Statistics Manual for Mental Disorders (DSM-5)

Exclusion Criteria:

* If participants report a history of psychiatric disorders within the past 12 months such as schizophrenia, dementia, depression, alcohol and other drug addiction.
* Participants could not partake if they were pregnant
* Participants enroll in another psychological treatment program.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Change: Social anxiety | a measure assessing change between three time points (pre-test, post-test (after two months), and follow-up test (after four months)
  Liebowitz Social Anxiety Scale for measuring social anxiety. this scale comprises of fear or anxiety and avoidance and sub-scales are combine (summed) to compute total score. Total score ranging from 0 to 144, and An individual who gets a total score over 60 in this measure is considered to have social anxiety

SECONDARY OUTCOMES:
Change: Rumination and Reflection | a measure assessing change between three time points (pre-test, post-test (after two months), and follow-up test (after four months))
  Rumination and Reflection Questionnair for measuring rumination and reflection: This scale comprises rumination and reflection. Each sub-scale comprises 12 items, and total scores ranged from 12 to 60. An individual who gets higher score is considered to have high rumination/ reflection.

OTHER OUTCOMES:
Change:Perfectionism | a measure assessing change between three time points (pre-test, post-test (after two months), and follow-up test (after four months)
  Almost Perfect Scale-Revised for measuring perfectionism: This scale comprises 23 items, but only 12 items associated to discrepancy (as a measure of maladaptive perfectionism or clinical perfectionism) are utilized in this study. Total scores ranged from 12 to 84 and higher score indicates higher level of perfectionism.

IPD SHARING:
Plan to Share IPD: Undecided